CLINICAL TRIAL: NCT06877923
Title: Evaluating the Tolerance, Compliance and Acceptability of a Nutritionally Complete Amino Acid-based Nutritional Supplement for the Dietary Management of Conditions With a Severe Impairment of the Gastrointestinal Tract in Children and Adults: a Case Study Series
Brief Title: Elemental 028 Extra Case Studies
Acronym: E028E
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E028E; 329442 (Other: IRAS)
Record Dates: First submitted 2025-02-21; First posted 2025-03-14 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Gastrointestinal Disease; Inflammatory Bowel Disease (IBD); Short Bowel; Malabsorption; Allergies; Neurodegenerative Disorders
MeSH Terms: conditions — Gastrointestinal Diseases; Inflammatory Bowel Diseases; Malabsorption Syndromes; Hypersensitivity; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elemental 028 Extra New Formulation (Experimental)
  Interventions: Dietary Supplement: Elemental 028 Extra

INTERVENTIONS:
Dietary Supplement: Elemental 028 Extra — Elemental 028 Extra formulations. Both powder and liquid versions will be used

SUMMARY:
Elemental 028 Extra is a nutritionally complete ACBS approved amino acid-based (elemental) feed designed to provide adequate daily amounts of both macronutrients and micronutrients when used as a sole source of nutrition and to support patients with severe impairment of the gastrointestinal tract who may require an elemental diet. An upgraded formulation of Elemental 028 Extra with an increased energy, protein content micronutrient profile has been developed to better meet the nutritional requirements of patients.

This series of case-studies aims to evaluate the acceptability, compliance, and gastrointestinal tolerance of the upgraded formulation of Elemental 028 Extra, in 30 adult and paediatric patients (15 powder and 15 liquid), with conditions where there is a severe impairment of the gastrointestinal tract, such as inflammatory bowel disease, short bowel syndrome, intractable malabsorption, allergic disease, and neurodegenerative diseases, and an elemental feed is required. The case study will last 29 days in total, including a 1-day baseline period followed by a 28-day intervention period. The case studies will be conducted across multiple centres in the UK, to meet the UK ACBS and GMS requirements for acceptability studies.

DETAILED DESCRIPTION:
Medical nutrition feeds for the dietary management of gastrointestinal impairment and/or allergic diseases can be broadly classified into three categories according to the size of the protein source in the feed: polymeric, extensively or partially hydrolysed, and elemental feeds. Polymeric feeds contain whole protein sources, typically from milk, soy, or pea protein. Extensively or partially hydrolysed feeds, also referred to as oligopeptide or semi-elemental feeds, contain peptides which are on average 4-5 amino acids in length, and are typically hypoallergenic as the peptides are too short for antigen recognition or presentation. Elemental feeds, also referred to as amino acid-based, hydrolysed or pre-digested, contain single amino acids as a source of protein and have a broad clinical application amongst patients with conditions where there is a severe impairment of the gastrointestinal tract possibly due to maldigestion and/or malabsorption including inflammation, reduced concentration of digestive enzymes and/or reduced surface area for nutrient absorption associated with some diseases and treatments. Such conditions include gastrointestinal diseases or disorders, neuro-disabilities and neuro-degenerative diseases, gynaecological cancers, and gastrointestinal impairment secondary to clinical treatment. Allergic diseases can also be managed with elemental feeds.

Elemental 028 Extra is a nutritionally complete ACBS approved amino acid-based (elemental) feed designed to provide adequate daily amounts of both macronutrients and micronutrients when used as a sole source of nutrition and to support patients with severe impairment of the gastrointestinal tract who may require an elemental diet. An upgraded formulation of Elemental 028 Extra with an increased energy, protein content and micronutrient profile has been developed to better meet the nutritional requirements of patients.

This series of case-studies aims to evaluate the acceptability, compliance, and gastrointestinal tolerance of the upgraded formulation of Elemental 028 Extra, in 30 adult and paediatric patients (15 powder and 15 liquid), with conditions where there is a severe impairment of the gastrointestinal tract, such as inflammatory bowel disease, short bowel syndrome, intractable malabsorption, allergic disease, and neurodegenerative diseases, and an elemental feed is required. The case study will last 29 days in total, including a 1-day baseline period followed by a 28-day intervention period. The case studies will be conducted across multiple centres in the UK, to meet the UK ACBS and GMS requirements for acceptability studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Over 3 years of age
* Requiring an elemental feed (at least 30% of total energy requirements)
* Written or electronic informed consent from patient, and/or from parent/caregiver if applicable

Exclusion Criteria:

* Pregnant or lactating
* Requiring parenteral nutrition
* Major hepatic or renal dysfunction
* Participation in other studies within 1 month prior to entry of this study
* Investigator concern around willingness/ability of patient or parent/caregiver to comply with protocol requirements

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Gastro-intestinal tolerance | Will be recorded at baseline (day 1) and end of intervention (day 29)
  Gastro-intestinal (GI) tolerance will be recorded by the Dietitian at baseline on Day 1 and at the end of the case study period. GI tolerance will be recorded using a standardised questionnaire (rating their symptoms from None, Mild, Moderate to Severe), to be completed by the patient or caregiver, as appropriate. Patients and/or parents/caregivers will be asked to record their symptoms in the past 24 hours and as an average over the case study period.

SECONDARY OUTCOMES:
Acceptability | Measured at baseline (day 1) and end of intervention period (day 29).
  Acceptability (ease of use and liking) of the patients' usual/current feed will be assessed by the Dietitian at baseline (Day 1) and of the study product at the end of the case study period by a series of questions posed to the patient and/or parent/caregiver. Acceptability questions will assess the patient's sensory experience, ease of use, tolerance, and overall self-rated acceptability on a 5-point Likert scale (rating from Great to Terrible).
Compliance | Measured at baseline (day 1) and end of intervention period (day 29).
  Compliance (volume and % of product consumed) with the prescribed intake of the patients' current feed(s) (before starting the intervention period) and with the study product (during the intervention period) will be assessed by the Dietitian at baseline (Day 1) and at the end of the case study period, respectively. Patients and/or parents/caregivers will be asked to recall the volume of feed consumed in the past 24 hours and on average. This will be compared to the amount recommended to consume by their Dietitian. The daily amount prescribed by the Dietitian managing the patient's care will be recorded at the start of the case study and any changes to this prescription during the case study will also be noted
Anthropometry | Measured at baseline (day 1) and end of intervention period (day 29).
  For safety purposes, at baseline (Day 1) and at the end of the case study, body weight (kg) will be measured where possible using standard methods, recorded to the nearest 0.1kg using a weighing scale without heavy clothing. Height will also be measured, using standard methods, recorded to the nearest 0.1cm (at baseline only) and used to calculate body mass index (BMI, kg/m2).

OTHER OUTCOMES:
Patient history | Measured at baseline only.
  A detailed patient history will be recorded at baseline to assess previously prescribed nutrition feeds, relevant medical and clinical issues, medication(s) prescribed, and any other relevant information related to the patient's condition or dietary management.
Safety | Measured throughout the full study period. From day 1 through to day 29.
  All adverse events will be recorded, throughout the case study.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hubbard, Study Director — Nutricia UK